CLINICAL TRIAL: NCT06582641
Title: Evaluation of Peer Group Connection - Middle School (PGC-MS)
Brief Title: Evaluation of Peer Group Connection - Middle School
Acronym: PGC-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Mathematica Policy Research, Inc. (Other); Reproductive Health National Training Center (Unknown); Center for Supportive Schools (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1 TP2AH000083-01-00
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer Group Connection - Middle School (PGC-MS) (Experimental)
  Interventions: Behavioral: Peer Group Connection - Middle School (PGC-MS)
- Class as usual (No Intervention)

INTERVENTIONS:
Behavioral: Peer Group Connection - Middle School (PGC-MS) — Peer Group Connection - Middle School (PGC-MS) is the treatment condition. PGC-MS is a school-based positive youth development program for students entering the transition year into middle school (6th or 7th grade). PGC-MS aims to improve school engagement and social-emotional learning skills that support adolescent health and educational outcomes for program participants. Participants receive 45-minute outreach sessions held 3 to 4 times per month for the full school year. Schools are expected to implement a minimum of 18 outreach sessions over the school year. PGC-MS outreach sessions are delivered by older peer leaders (8th, 9th, or 10th graders) who are carefully selected by faculty advisors and trained on how to deliver program content.
  Arms: Peer Group Connection - Middle School (PGC-MS)

SUMMARY:
The goal of this randomized trial is to learn if the Peer Group Connection - Middle School (PGC-MS) intervention delays initiation of sexual intercourse in middle school-aged youth. The primary research question it aims to answer is:

Sixteen months after being offered the intervention, does PGC-MS impact youth's initiation of sexual intercourse?

Researchers will compare participants randomized to receive PGC-MS (treatment group) to participants randomized to class-as-usual (which contains no sexual or reproductive health information (control group)).

Participants randomized to the treatment group will be offered PGC-MS over the course of their transition year into middle school (either 6th or 7th grade). Participants randomized to the control group will be offered class-as-usual.

DETAILED DESCRIPTION:
This is an individual-level, randomized control trial to rigorously evaluate the impact of the Peer Group Connection - Middle School (PGC-MS) intervention. Participant outcomes will be assessed using self-reported, individual-level data gathered using a structured questionnaire administered at four time points: baseline (fall semester of 6th or 7th grade); post-intervention (spring semester of 6th or 7th grade); four months post-intervention (fall semester of 7th or 8th grade); and sixteen months post-intervention (fall semester of 8th or 9th grade).

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled at a middle school participating in the study
* Entering the middle school transition grade for the first time (6th or 7th grade depending on the middle school transition year) at a participating study school
* Provide parental consent and student assent to participate in the study
* Have the ability to complete a self-administered questionnaire in either English or Spanish in a classroom or group setting, unassisted, in 60 minutes or less.

Exclusion Criteria:

- Repeating the middle school transition year (6th or 7th grade)

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1400 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
Initiation of sexual intercourse | Assessed 16 months after the intervention period has ended (beginning of the second fall semester following the end of the program)
  Participants are asked the following item: 1) Have you ever had sexual intercourse? The resulting variable is dichotomous with values 0 or 1, where 0 indicates a person who has never sexual intercourse and 1 indicates a person who has had sexual intercourse.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Walsh, PhD, Principal Investigator — The Policy & Research Group
Locations (1):
- The Policy & Research Group, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes de-identified individual-level data on all study participants who contributed self-report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program components were completed). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Supporting Information: SAP
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.